CLINICAL TRIAL: NCT01650519
Title: A Pilot Study to Determine the Efficacy of Intravenous Ibuprofen for Pain Control Following Arthroscopic Knee Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CPI-CL-017
Record Dates: First submitted 2012-07-24; First posted 2012-07-26 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Arthroscopic Knee Surgery
Keywords: knee surgery, arthroscopy; orthopaedic, orthopedic surgery
MeSH Terms: interventions — Ibuprofen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV ibuprofen (Active Comparator): Intravenous ibuprofen (800 mg) administered intravenously over 10 minutes at study hour 0 and again at study hour 4 (Ibuprofen arm) and a corresponding volume of normal saline (ketorolac arm) will be administered intravenously over no less than 15 seconds at the end of the arthroscopic procedure
  Interventions: Drug: IV ibuprofen
- IV ketorolac (Active Comparator): A corresponding volume of normal saline (Ibuprofen arm) administered intravenously over 10 minutes at study hour 0 and again at study hour 4 and 30 mg ketorolac for patients < 65 years of age (15 mg ketorolac for patients > 65 years of age) (ketorolac arm) will be administered intravenously over no less than 15 seconds at the end of the arthroscopic procedure
  Interventions: Drug: IV ketorolac

INTERVENTIONS:
Drug: IV ibuprofen — 800 mg intravenous ibuprofen administered intravenously over 10 minutes.
  Other Names: Caldolor
  Arms: IV ibuprofen
Drug: IV ketorolac — 30 mg ketorolac for patients < 65 years of age (15 mg ketorolac for patients > 65 years of age) administered intravenously over no less than 15 seconds
  Other Names: Toradol
  Arms: IV ketorolac

SUMMARY:
The intent of this study is to assess the analgesic efficacy of IV ibuprofen when administered at induction of anesthesia. Results from this pilot study will be used to design and determine the appropriate statistical power for a larger, multi-center randomized study.

DETAILED DESCRIPTION:
Non-steroidal anti-inflammatory drugs(NSAIDs) are an effective adjunct to opioid analgesia for moderate-severe pain, with improvement in the quality of pain relief and consistent evidence of opioid dose sparing. NSAIDs alone could provide effective analgesia post-surgery when mild-moderate pain is expected. There is also evidence that the use of NSAIDs, by avoiding or decreasing the need for opioids, can lead to a reduction in the incidence of adverse events which are commonly attributed to, or exacerbated by, opioids.

The intent of this study is to assess the analgesic efficacy of IV ibuprofen when administered at induction of anesthesia. Results from this pilot study will be used to design and determine the appropriate statistical power for a larger, multi-center randomized study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for knee arthroscopy

Exclusion Criteria:

* Inadequate intravenous (IV) access.
* History of allergy or hypersensitivity to any component of ibuprofen or other NSAIDs, aspirin (or aspirin related products), opioids or cyclooxygenase-2(COX-2) inhibitors.
* Less than 18 years of age.
* Use of analgesics less than 8 hours prior to surgery.
* Patients with active, clinically significant anemia.
* History or evidence of asthma or heart failure.
* Pregnant.
* Recent history of chronic non-steroidal anti-inflammatory drug (NSAID) or opioid use.
* Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions and to return for the required assessments.
* Refusal to provide written authorization for use and disclosure of protected health information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando L Arbona, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Wexner Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Uribe AA, Arbona FL, Flanigan DC, Kaeding CC, Palettas M, Bergese SD. Comparing the Efficacy of IV Ibuprofen and Ketorolac in the Management of Postoperative Pain Following Arthroscopic Knee Surgery. A Randomized Double-Blind Active Comparator Pilot Study. Front Surg. 2018 Oct 3;5:59. doi: 10.3389/fsurg.2018.00059. eCollection 2018. PMID 30338261

RESULTS

PARTICIPANT FLOW:
Groups:
- IV Ibuprofen: 800 mg intravenous ibuprofen administered intravenously over 10 minutes at hour 0 and again at hour 4. 30 mg NS < 65 years of age (15 mg NS for patients > 65 years of age) administered intravenously over no less than 15 seconds at reversal of anesthesia.
  IV ibuprofen: 800 mg intravenous ibuprofen administered intravenously over 10 minutes.
- IV Ketorolac: Either 30 mg ketorolac for patients < 65 years of age (15 mg ketorolac for patients > 65 years of age) administered intravenously over no less than 15 seconds at reversal of anesthesia. 800 mg NS administered intravenously over 10 minutes at hour 0 and hour 4.
  IV ketorolac: 30 mg ketorolac for patients < 65 years of age (15 mg ketorolac for patients > 65 years of age) administered intravenously over no less than 15 seconds
Period: Overall Study
Arm/Group | IV Ibuprofen | IV Ketorolac
Started | 20 | 31
Completed | 19 | 31
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat population consists of all patients who received at least a partial dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | IV Ibuprofen | IV Ketorolac | Total
Number analyzed (Participants) | 20 | 31 | 51
Age, Customized [Mean (Standard Deviation); unit: years] — Subject greater than or equal to 18 years of age
  years
    Subject greater than or equal to 18 years of age | 43 (12.6) | 45 (13) | 44 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 14 | 21 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 17 | 29 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 30 | 50
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 31 | 51

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of IV Ibuprofen for Post-op Pain.
Description: Measurement of the efficacy of IV ibuprofen for the treatment of postoperative pain as measured by patient pain intensity (Visual Analog Scale, VAS) upon first possible assessment following surgery. The VAS is a continuous scale compromised of a horizontal line, one hundred millimeters in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between o and 100.
Time Frame: first possible assessment following surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Ibuprofen | IV Ketorolac
Number analyzed (Participants) | 19 | 31
units on a scale
  VAS at Rest (mm) | 8 (6.6) | 34 (25.0)
  VAS with Movement (mm) | 19 (17.4) | 41 (25.8)

2. Secondary Outcome: Measurement of the Efficacy of IV Ibuprofen for the Treatment of Postoperative Pain as Measured by the Amount of Rescue Medication in the Postoperative Period Through Discharge
Description: Measurement of the amount of rescue medication in the postoperative period.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | IV Ibuprofen | IV Ketorolac
Number analyzed (Participants) | 19 | 31
milligrams
  Narcotic | 5.4 (6.02) | 20.4 (15.87)
  Acetaminophen | 162.5 (229.81) | 325 (269.90)

3. Secondary Outcome: Time to Discharge.
Description: Measurement of the time to discharge in the postoperative period.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV Ibuprofen | IV Ketorolac
Number analyzed (Participants) | 19 | 31
Hours | 1.8 (0.12) | 1.8 (0.08)

4. Secondary Outcome: Patient Satisfaction.
Description: Measurement of patient satisfaction post-procedure. During the post-treatment period, subjects were asked to complete a satisfaction questionnaire (Quality of Recovery - 40 or QoR-40) defining their quality of recovery at 24 hours following surgery. The QoR - 40 is a 40-item questionnaire that provides a global score and subscores across five dimensions of quality of recovery: emotions (minimum score = 6, maximum score = 30), physical comfort (minimum score = 8, maximum score = 40), patient support (minimum score = 7, maximum score = 35), physical independence (minimum score = 5, maximum score = 25), and pain (minimum score = 7, maximum score = 35). Higher subscores represent a better outcome.
  Subscores are added to create a Global QoR-40 score. Global scores range from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IV Ibuprofen | IV Ketorolac
Number analyzed (Participants) | 13 | 18
units on a scale
  Emotions | 20.2 (2.35) | 20.7 (2.25)
  Physical Comfort | 28.3 (4.39) | 26.9 (2.98)
  Patient Support | 30.5 (1.20) | 29.0 (3.93)
  Physical Independence | 22.2 (2.55) | 21.3 (3.32)
  Pain | 9.5 (3.45) | 10.9 (3.34)

5. Secondary Outcome: Incidence of Serious Adverse Events (SAEs).
Description: Measurement of the incidence of serious adverse events.
Time Frame: 24 hours
Measure: Number; unit: Number of Events
Arm/Group | IV Ibuprofen | IV Ketorolac
Number analyzed (Participants) | 20 | 31
Number of Events | 0 | 0

6. Secondary Outcome: Measurement of the Efficacy of IV Ibuprofen for the Treatment of Postoperative Pain as Measured by the Pain Intensity as Assess by Patient Pain Intensity (VAS) in the Post-surgical Period, Through 24 Hours
Description: Measurement of the efficacy of IV ibuprofen for the treatment of postoperative pain as measured by patient pain intensity (Visual Analog Scale, VAS) in the post-surgical period through 24 hours post-procedure. The VAS is a continuous scale made up of a horizontal line, 100 mm in length, anchored by 2 verbal descriptors (No Pain, Worst Possible Pain). The VAS is self-completed by the respondent. The subject is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. Using a ruler, the score is determined by measuring the distance, in mm, on the 100 mm line between the "No Pain" anchor and the subject's mark. The score would be between 0 and 100. Subject's were contacted at 24 hour post-discharge during a follow-up phone contact and asked to completed the VAS at Rest and VAS with Movement and return both completed VAS assessments via the envelope provided. The analysis was performed on the VAS assessments returned to the study site.
Time Frame: 24 Hours
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | IV Ibuprofen | IV Ketorolac
Number analyzed (Participants) | 10 | 13
units on a scale
  VAS at Rest (mm) | 4 (3.7) | 13 (10.8)
  VAS with Movement (mm) | 12 (12.2) | 23 (16.5)

7. Secondary Outcome: Measurement of the Efficacy of IV Ibuprofen for the Treatment of Postoperative Pain as Measured by the Amount of Time to Rescue Medication in the Postoperative Period Through Discharge
Description: Measurement of the amount of time to rescue medication in the postoperative period.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | IV Ibuprofen | IV Ketorolac
Number analyzed (Participants) | 20 | 31
Hours | 1.7 (0.19) | 1 (0.11)

ADVERSE EVENTS:
Arm/Group | IV Ibuprofen | IV Ketorolac
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/31
Other Adverse Events (participants affected / at risk) | 0/20 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No